CLINICAL TRIAL: NCT00002798
Title: A PHASE III STUDY IN CHILDREN WITH UNTREATED ACUTE MYELOGENOUS LEUKEMIA (AML) OR MYELODYSPLASTIC SYNDROME (MDS)
Brief Title: Combination Chemotherapy With or Without Bone Marrow Transplantation in Treating Children With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01834; 2961; U10CA098543 (NIH); CDR0000064883 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-11-24; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myelomonocytic Leukemia (M4); Childhood Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Anemia With Ringed Sideroblasts; Secondary Myelodysplastic Syndromes; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Asparaginase; palmitoyl-L-asparaginase; Daunorubicin; fludarabine phosphate; Hydrocortisone; Transplantation; Radiotherapy, Conformal; Filgrastim; Granulocyte Colony-Stimulating Factor; Cytarabine; Idarubicin; Dexamethasone; Calcium Dobesilate; Thioguanine; Etoposide; Methotrexate; merphos; Cyclophosphamide; aldesleukin; Interleukin-2; Busulfan

ARMS (5):
- Arm I (combination chemotherapy) (Experimental): Patients receive treatment as in induction therapy, plus G-CSF SC beginning on day 16 and continuing until blood counts recover. If CSF is clear by day 10 of induction, patients receive cytarabine IT on days 0, 10, and 35. If CSF is not clear, patients receive triple intrathecal therapy (TIT; cytarabine, hydrocortisone, methotrexate) on days 0 and 10.
  See Detailed Description
  Interventions: Drug: daunorubicin hydrochloride; Drug: therapeutic hydrocortisone; Procedure: allogeneic bone marrow transplantation; Biological: filgrastim; Drug: cytarabine; Drug: idarubicin; Drug: dexamethasone; Drug: thioguanine; Drug: etoposide; Drug: methotrexate
- Arm II (combination chemotherapy) (Experimental): Patients receive fludarabine IV over 24 hours on days 0 and 1, cytarabine IV over 72 hours on days 2-4, and idarubicin IV over 15 minutes on days 0-2. G-CSF begins on day 6 and continues until blood counts recover. Patients also receive TIT on days -1 and 7, if CSF is not clear on day 10 of induction. Patients on both arms are reassessed on day 35. Those patients with M1 marrow proceed to intensification; all others are removed from the study.
  Intensification: See Detailed Description
  Interventions: Drug: asparaginase; Drug: fludarabine phosphate; Drug: therapeutic hydrocortisone; Procedure: allogeneic bone marrow transplantation; Biological: filgrastim; Drug: cytarabine; Drug: idarubicin; Drug: thioguanine; Drug: methotrexate; Drug: cyclophosphamide; Drug: busulfan
- Arm III (combination chemotherapy, aldesleukin) (Experimental): Patients receive interleukin-2 IV continuously on days 1-4 and 9-18.
  Interventions: Drug: daunorubicin hydrochloride; Biological: filgrastim; Drug: cytarabine; Drug: idarubicin; Drug: dexamethasone; Drug: thioguanine; Drug: etoposide; Biological: aldesleukin
- Arm IV (combination chemotherapy) (Active Comparator): No further treatment
  Interventions: Drug: daunorubicin hydrochloride; Biological: filgrastim; Drug: cytarabine; Drug: idarubicin; Drug: dexamethasone; Drug: thioguanine; Drug: etoposide
- Arm V (combination chemotherapy, radiotherapy) (Experimental): Patients undergo radiotherapy to the chloroma 5 days a week for 2 weeks.
  Interventions: Drug: daunorubicin hydrochloride; Radiation: 3-dimensional conformal radiation therapy; Biological: filgrastim; Drug: cytarabine; Drug: idarubicin; Drug: dexamethasone; Drug: thioguanine; Drug: etoposide

INTERVENTIONS:
Drug: asparaginase
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
  Arms: Arm II (combination chemotherapy)
Drug: daunorubicin hydrochloride
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
  Arms: Arm I (combination chemotherapy); Arm III (combination chemotherapy, aldesleukin); Arm IV (combination chemotherapy); Arm V (combination chemotherapy, radiotherapy)
Drug: fludarabine phosphate
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
  Arms: Arm II (combination chemotherapy)
Drug: therapeutic hydrocortisone
  Other Names: Aeroseb-HC; Barseb HC; Cetacort; Cort-Dome; Cortef
  Arms: Arm I (combination chemotherapy); Arm II (combination chemotherapy)
Procedure: allogeneic bone marrow transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
  Arms: Arm I (combination chemotherapy); Arm II (combination chemotherapy)
Radiation: 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
  Arms: Arm V (combination chemotherapy, radiotherapy)
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Drug: cytarabine — Given IV or IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
  Arms: Arm I (combination chemotherapy); Arm III (combination chemotherapy, aldesleukin); Arm IV (combination chemotherapy); Arm V (combination chemotherapy, radiotherapy)
Drug: thioguanine — Given PO
  Other Names: 6-TG
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Arm I (combination chemotherapy); Arm III (combination chemotherapy, aldesleukin); Arm IV (combination chemotherapy); Arm V (combination chemotherapy, radiotherapy)
Drug: methotrexate — Given IT
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
  Arms: Arm I (combination chemotherapy); Arm II (combination chemotherapy)
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Arm II (combination chemotherapy)
Biological: aldesleukin
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
  Arms: Arm III (combination chemotherapy, aldesleukin)
Drug: busulfan
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
  Arms: Arm II (combination chemotherapy)

SUMMARY:
Randomized phase III trial to compare the effectiveness of different chemotherapy regimens with or without bone marrow transplantation in treating children who have acute myelogenous leukemia or myelodysplastic syndrome. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. It is not yet known which treatment regimen is more effective for acute myelogenous leukemia or myelodysplastic syndrome

DETAILED DESCRIPTION:
OBJECTIVES:

Increase the remission induction rate to greater than 85% in children with untreated acute myelogenous leukemia (AML) or myelodysplastic syndromes (MDS) by replacing daunorubicin (DNR) with idarubicin (IDA) in intensively timed DCTER chemotherapy (dexamethasone, cytarabine (ARA-C), thioguanine, etoposide, and daunorubicin) in the first 4 days of each course.

Increase the remission rate further by comparing the efficacy of consolidation chemotherapy with intensively timed IDA DCTER/DCTER vs fludarabine (FAMP), ARA-C, and IDA in maintaining remission and in achieving remission in patients with M2 disease (5%-29% blasts in marrow) at the end of induction chemotherapy.

Compare overall survival, event-free survival, and disease-free survival in patients who receive consolidation with IDA DCTER/DCTER vs FAMP, ARA-C, and IDA.

Compare overall survival, event-free survival, and disease-free survival in patients receiving intensification with the Capizzi II regimen (high-dose ARA-C and asparaginase) vs those receiving a matched-related allogeneic bone marrow transplantation.

Compare overall survival, event-free survival, and disease-free survival in patients treated with interleukin-2 (IL-2) vs standard follow up care after Capizzi II intensification.

Determine whether multichannel flow cytometry detection of residual AML on a companion biologic study protocol CCG-B942 predicts outcome, and determine whether any of these treatment regimens eliminates minimal residual disease more effectively than another.

Register all patients with MDS treated or followed at CCG institutions and capture their biologic, historical and outcome data.

Determine, on a companion biologic study protocol CCG-B972, whether levels of IL-2 soluble receptor (sIL-2R) and absolute lymphocyte count (ALC) before, during, and after therapy correlates with outcome.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, diagnosis (acute myelogenous leukemia vs other), and response to induction (partial vs complete remission). After induction, patients with M1/M2 marrow are randomized to arm I or II. Patients in complete remission after consolidation who have an HLA-identical or 1-antigen mismatched sibling or parent donor are randomly assigned to the allogeneic bone marrow transplantation (AlBMT) regimen; all others in complete remission are nonrandomly assigned to the Capizzi II regimen, then are randomly assigned to arms III or IV. Patients with refractory anemia (RA) or RA with ringed sideroblasts with indolent disease may be registered and followed. Other patients with myelodysplastic syndromes may receive 2961 chemotherapy or go directly to AlBMT. Patients with chloromas (granulocytic sarcomas) receive optional radiotherapy on arm V.

Induction: Patients receive idarubicin IV over 30 minutes on days 0-3, cytarabine and etoposide IV continuously on days 0-3, and oral thioguanine twice a day and oral dexamethasone 3 times a day on days 0-3. Patients then begin course 2, which consists of cytarabine, etoposide, thioguanine, and dexamethasone on days 10-13, daunorubicin IV continuously on days 10-13, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 16 and continuing until blood counts recover. Patients also receive CNS prophylaxis/therapy consisting of cytarabine intrathecally (IT) on days 0 and 14 (if no CNS disease at entry) or on days 0, 5, and 7 (if CNS disease present at entry). Disease is reassessed on day 28-42. Patients with M1 or M2 marrow proceed to consolidation while those with M3 marrow or progressive disease go off study.

Consolidation:

Arm I: Patients receive treatment as in induction therapy, plus G-CSF SC beginning on day 16 and continuing until blood counts recover. If CSF is clear by day 10 of induction, patients receive cytarabine IT on days 0, 10, and 35. If CSF is not clear, patients receive triple intrathecal therapy (TIT; cytarabine, hydrocortisone, methotrexate) on days 0 and 10.

Arm II: Patients receive fludarabine IV over 24 hours on days 0 and 1, cytarabine IV over 72 hours on days 2-4, and idarubicin IV over 15 minutes on days 0-2. G-CSF begins on day 6 and continues until blood counts recover. Patients also receive TIT on days -1 and 7, if CSF is not clear on day 10 of induction. Patients on both arms are reassessed on day 35. Those patients with M1 marrow proceed to intensification; all others are removed from the study.

Intensification:

Capizzi II regimen: Course 1: Patients receive cytarabine IV over 3 hours every 12 hours on days 0, 1, 7, and 8 and asparaginase IM on days 1 and 8. Course 2: Patients also receive cytarabine IT or TIT on days 0, 7, and 14.AlBMT regimen: Therapy begins within 2-8 weeks of hematologic recovery. Patients may receive interim therapy consisting of oral thioguanine for about 2 weeks. Patients then receive oral busulfan every 6 hours on days -9 to -6 and cyclophosphamide IV over 1 hour on days -5 to -2. AlBMT is infused over 4 hours beginning 36-48 hours after the last dose of cyclophosphamide. Patients in complete remission after completing the Capizzi II regimen proceed to maintenance therapy on arm III.

Arm III: Patients receive interleukin-2 IV continuously on days 1-4 and 9-18.

Arm IV: No further treatment.

Arm V: Patients undergo radiotherapy to the chloroma 5 days a week for 2 weeks.

Patients are followed monthly for 18 months, every 3 months for 1 year, and then every 6 months until 5 years from diagnosis.

PROJECTED ACCRUAL: Approximately 880 patients with de novo acute myelogenous leukemia will be accrued for this study within 4 years. It is expected that 178 patients per year will be randomly assigned for consolidation, that 39 patients per year will undergo allogeneic bone marrow transplantation while 120 patients per year will receive chemotherapy as intensification, and that 102 patients per year will be randomly assigned for polychemotherapy immunomodulation. An additional 80 patients with myelodysplastic syndromes will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed previously untreated acute myeloid leukemia (AML) in patients 1 month to 21 years of age

  * Infants under 1 month with progressive disease eligible

    * Supportive care may be given to confirm that the leukemia is not regressing prior to entry
  * No acute promyelocytic leukemia (FAB M3)
  * No acute undifferentiated leukemia (FAB M0)
* Histochemical verification of AML required by the following stains:

  * Wright or Giemsa
  * Peroxidase
  * PAS
  * Chloroacetate esterase
  * Sudan black
  * Nonspecific esterase (NSE) with and without fluoride (NaF) inhibition
  * Combined NSE/NaF and butyrate inhibition or diagnosis of megakaryoblasticleukemia (FAB M7) should be supported by one of the following:

    * CD41 reactivity
    * Glycoprotein 1b reactivity
    * Factor VIII-related antigen reactivity
    * Platelet peroxidase on electron microscopy
* The following are also eligible:

  * Myelodysplastic syndromes, including:

    * Refractory anemia (RA) *
    * RA with ringed sideroblasts (RARS) *
    * RA with excess blasts (RAEB)
    * RAEB in transformation (RAEBt)
    * Chronic myelomonocytic leukemia (CMML)
  * AML with monosomy 7
  * Granulocytic sarcoma (chloroma) with or without marrow involvement
  * Mixed lineage leukemia with 2 morphologically defined populations provided the predominant population is myeloid
* No Downs syndrome
* No juvenile chronic myelogenous leukemia
* No Fanconi's anemia
* No secondary AML
* Performance status - Not specified
* No prior anticancer chemotherapy
* Prior topical or inhaled steroids for nonmalignant conditions allowed
* No prior anticancer radiotherapy
* No prior antileukemic therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 880 (Actual)
Dates: Start 1996-08; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Proportions of patients achieving remission rate during induction therapy | Up to 42 days
Proportion of patients dying or with residual disease during induction therapy | Up to 42 days
Time to marrow recovery (induction phase) | Up to 42 days
Frequency of toxicities, including infectious complications (induction phase) | Up to 42 days
Marrow status | At 14 days
Percent of blasts | At the end of induction therapy
Complete remission at the end of consolidation therapy | Up to 5 years
Survival following consolidation | Up to 5 years
Event-free survival following consolidation | Up to 5 years
Overall survival (intensification) | Up to 5 years
EFS (intensification) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Lange, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Derived] Tarlock K, Gerbing RB, Ries RE, Smith JL, Leonti A, Huang BJ, Kirkey D, Robinson L, Peplinski JH, Lange B, Cooper TM, Gamis AS, Kolb EA, Aplenc R, Pollard JA, Alonzo TA, Meshinchi S. Prognostic impact of cooccurring mutations in FLT3-ITD pediatric acute myeloid leukemia. Blood Adv. 2024 May 14;8(9):2094-2103. doi: 10.1182/bloodadvances.2023011980. PMID 38295280
- [Derived] Bertrums EJM, Smith JL, Harmon L, Ries RE, Wang YJ, Alonzo TA, Menssen AJ, Chisholm KM, Leonti AR, Tarlock K, Ostronoff F, Pogosova-Agadjanyan EL, Kaspers GJL, Hasle H, Dworzak M, Walter C, Muhlegger N, Morerio C, Pardo L, Hirsch B, Raimondi S, Cooper TM, Aplenc R, Gamis AS, Kolb EA, Farrar JE, Stirewalt D, Ma X, Shaw TI, Furlan SN, Brodersen LE, Loken MR, Van den Heuvel-Eibrink MM, Zwaan CM, Triche TJ, Goemans BF, Meshinchi S. Comprehensive molecular and clinical characterization of NUP98 fusions in pediatric acute myeloid leukemia. Haematologica. 2023 Aug 1;108(8):2044-2058. doi: 10.3324/haematol.2022.281653. PMID 36815378
- [Derived] Ho PA, Zeng R, Alonzo TA, Gerbing RB, Miller KL, Pollard JA, Stirewalt DL, Heerema NA, Raimondi SC, Hirsch B, Franklin JL, Lange B, Meshinchi S. Prevalence and prognostic implications of WT1 mutations in pediatric acute myeloid leukemia (AML): a report from the Children's Oncology Group. Blood. 2010 Aug 5;116(5):702-10. doi: 10.1182/blood-2010-02-268953. Epub 2010 Apr 22. PMID 20413658
- [Derived] Pollard JA, Alonzo TA, Gerbing RB, Ho PA, Zeng R, Ravindranath Y, Dahl G, Lacayo NJ, Becton D, Chang M, Weinstein HJ, Hirsch B, Raimondi SC, Heerema NA, Woods WG, Lange BJ, Hurwitz C, Arceci RJ, Radich JP, Bernstein ID, Heinrich MC, Meshinchi S. Prevalence and prognostic significance of KIT mutations in pediatric patients with core binding factor AML enrolled on serial pediatric cooperative trials for de novo AML. Blood. 2010 Mar 25;115(12):2372-9. doi: 10.1182/blood-2009-09-241075. Epub 2010 Jan 7. PMID 20056794
- [Derived] Ho PA, Alonzo TA, Gerbing RB, Pollard J, Stirewalt DL, Hurwitz C, Heerema NA, Hirsch B, Raimondi SC, Lange B, Franklin JL, Radich JP, Meshinchi S. Prevalence and prognostic implications of CEBPA mutations in pediatric acute myeloid leukemia (AML): a report from the Children's Oncology Group. Blood. 2009 Jun 25;113(26):6558-66. doi: 10.1182/blood-2008-10-184747. Epub 2009 Mar 20. PMID 19304957